CLINICAL TRIAL: NCT01548209
Title: Effects of a Single Dose Dexmedetomidine on Postoperative Nausea and Vomiting (PONV) and Quality of Recovery 40 (QoR 40) in Breast Cancer Surgery
Brief Title: Effects of a Dexmedetomidine on Quality of Recovery 40 and Postoperative Nausea and Vomiting in Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2011-0415
Record Dates: First submitted 2012-02-27; First posted 2012-03-08 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group D (Experimental): A single dose dexmedetomidine 0.5 mcg/kg iv. 30 min before end of the surgery
  Interventions: Drug: Dexmedetomidine
- Group P (Placebo Comparator): Placebo 0.5 mcg/kg iv. 30 min before end of the surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — A single dose dexmedetomidine 0.5 mcg/kg IV. 30 min before end of the surgery
  Arms: Group D
Drug: Placebo — Placebo 0.5 mcg/kg iv. 30 min before end of the surgery
  Arms: Group P

SUMMARY:
Postoperative nausea and vomiting (PONV) is common following beast surgery. Dexmedetomidine was reported to a reduced PONV due to opioid-sparing effect. It is not clear if dexmedetomidine itself is useful on reducing PONV. The hypothesis of present study: intraoperative application of single dose dexmedetomidine (0.5 mcg/kg) is is effective than placebo for reducing of PONV and improve postoperative quality of recovery score within 48 postoperative hours.

DETAILED DESCRIPTION:
This study was approved by the Institutional Review Board of Severance Hospital, Yonsei University Health System. After written informed consent was obtained from all patients, aged 20-75 years with ASA physical status class I-II who were scheduled breast cancer surgery under general anaesthesia were enrolled in this study All the patients were randomly assigned to receive dexmedetomidine or placebo during surgery. The primary outcome was quality of recovery determined by QOR-40 in the first 24h after surgery.The secondary outcome measure was PONV assessed by visual analogue scale every 6 hours within 48 postoperative hours.

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II
* aged 20-70 years
* Undergoing breast cancer surgery

Exclusion Criteria:

* CAOD
* Bradycardia
* QT prolongation

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2011-09; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery 40 (QoR-40) | 24 postoperative hours
  quality of recovery was determined by QOR-40 questionnaire.
  (all same as Dexmedetomidine group and Placebo group)

SECONDARY OUTCOMES:
Change from preoperative baseline in PONV within 48 postoperative hours | every 6 hours within 48 postoperative hours
  PONV was determined by visual analogue scale, number of emetic episode every 6 hours within 48 postoperative hours
  (all same as Dexmedetomidine group and Placebo group)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, 250 Seungsan-no, Seodaemun-gu, Seoul, South Korea